CLINICAL TRIAL: NCT02480036
Title: Combining Intraoperative Radiotherapy With Kyphoplasty for Treatment of Spinal Metastases
Acronym: KYPHO-IORT
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Abhishek A. Solanki, Assistant Professor, Loyola University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 206824; 206824091714 (Other: Loyola University Chicago)
Record Dates: First submitted 2015-06-10; First posted 2015-06-24 (Estimated); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Spinal Metastasis
Keywords: IORT; Kyphoplasty; Spine; Cancer
MeSH Terms: conditions — Neoplasms | interventions — Kyphoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combined IORT and Kyphoplasty (Experimental): IORT with Kyphoplasty IORT Device: Intrabeam®
  Interventions: Radiation: IORT with Kyphoplasty; Device: Intrabeam®

INTERVENTIONS:
Radiation: IORT with Kyphoplasty — IORT with kyphoplasty is give concurrently for the treatment of spinal metastases
Device: Intrabeam®

SUMMARY:
The primary objective is to evaluate the tolerability (side effects) of the intraoperative radio therapy (IORT) (e.g., wound healing, infections, bone necrosis, nerve, spinal cord damage, and pathological fracture), and the secondary objective is to evaluate the effectiveness of IORT (i.e., pain relief, quality of life, narcotic use, and tumor response).

DETAILED DESCRIPTION:
Disease Background:

Bone metastases are the third most common site of metastatic spread, affecting 10% - 30% of all cancer patients. The spine remains the most common site of bone metastases, with incidence ranging from 30-70% depending on the primary tumour.

Spinal metastases can be a significant cause of morbidity for cancer patients: severe pain, bone fracture, nerve root or spinal cord compression, hypercalcemia, and limited mobility. Symptomatic spinal metastases are most frequently located in the thoracic spine (70%), followed by lumbar spine (20%) and cervical spine (10%). Up to 15% of all cancer patients with bone metastasis will suffer compression fracture leading to loss of function and the impairment of mobility, while more than 70% of the patients will experience severe cancer-related pain affecting quality of life. Newer systemic agents targeting specific pathway or molecule within the tumor milieu has led to a dramatic improvement in life expectancy for metastatic patients. Hence, effective palliative treatment options for spinal metastases is an important clinical issue in today's oncologic practice.

Current Practice:

The majority of patients with spinal metastases are initially managed medically with combination of analgesic medication, bisphosphonates, or biologic/chemotherapy agents.

When these patients develop severe pain refractory to medical options or there is a concern for neurologic dysfunction (i.e. vertebrate fracture, nerve root compression), they will be referred for palliative radiotherapy or surgical treatment options.

In the past decade, minimally invasive interventional therapies have become more popular to treat severe pain from spinal metastases, especially in patients with evidence of compression fracture. Vertebroplasty involves the percutaneous injection of cement into the vertebral body with the goals of pain alleviation and preventing further loss of vertebral body height. Similarly, in kyphoplasty (KYPHO), an inflatable balloon is used to create a cavity for the cement deposition, which restores height as well as provides pain relief. However, the immediate goal for both procedures is to achieve stabilization of the vertebral body and prevent further compression.

Investigators assessed the safety and efficacy of vertebroplasty and kyphoplasty for pain palliation in cancer patients. They performed ninety-seven procedures in fifty-six patients. The median age was 62 years. The procedure was well-tolerated and no post-operative complications or death were noted. There was a significant reduction in visual analog pain score (VAS): median pre-and postoperative VAS score was 7 and 2, respectively (P=0.001, student paired t-test). However, there concern for use of kyphoplasty alone in treatment of spinal metastases: the rate of re-treatment and variable duration of pain palliation. The rate of new compression fracture after balloon kyphoplasty in patients with malignant spinal fracture can be as high as 10%.

Non-surgical option to treat spinal metastases usually involves the use of external beam radiotherapy. The goals of radiation therapy are to alleviate pain, stabilize affected bone, and decrease tumor cells within the treated site. Radiotherapy is very effective in pain reduction, as 50-80% of all patients receiving palliative radiation will experience pain reduction. Pain reduction from ionizing radiation, in theory, is due to the direct analgesic effect on the nociceptors in the periosteum and electrolyte shift, which can convert pain-inducing tissue acidosis to tissue alkalosis. Furthermore, stabilization of the vertebral bodies can be achieved by decreasing number of tumor cells and hence, thereby changing the imbalance of osteoclast and osteoblast activity. The latter effect can increase re-mineralization. These effects will occur in 40-50% of patients after radiation therapy, but can take 4-6 weeks after external beam radiation therapy course.

Several issues arise with use of external beam radiation therapy. First, an optimal dose fraction schedule has not been well- established. The most common prescribed dose is 30 grays (Gy) in ten fractions. However, in Radiation Therapy Oncology Group (RTOG) 9714, investigators found no difference between 8Gy in single fraction versus extended 30Gy in 10 fraction schedule in terms of pain relief and narcotic medication usage at three months. Furthermore, an extended radiotherapy course can lead to patient inconvenience, longer hospitalization, and increased toxicity. In the RTOG 9714 trial, patients in the 30-Gy arm had more grade 2-4 toxicities than 8-Gy arm. Furthermore, there is a risk of vertebral fracture for patients treated with radiation therapy for spinal metastases. Researchers reported 31% of their patients with spinal cord compression treated with radiotherapy alone had vertebral collapse.

Hence, to achieve an optimal treatment option for symptomatic cancer patients with spinal metastases, the next logical step would be to combine stabilization (kyphoplasty) technique with direct tumor cell destruction in order to achieve maximum and durable pain palliation, prevent potential neurological dysfunction, and improve quality of life. By combining kyphoplasty with intraoperative radiation, one can achieve the above mentioned goals in a single outpatient procedure.

Combination of Kyphoplasty and Intraoperative Radiation:

During a surgical procedure, the tumor bed and/or the tumor itself can be irradiated with a single dose of radiation. Intraoperative radiation therapy [IORT] is the delivery of radiation during a surgical intervention. The advantages of the IORT consist of the high precision combined with optimal protection of the surrounding organs at risk. Hence, a higher dose of radiation can be applied to the target (as compared to external beam), while minimizing the adverse side effects to normal tissue. Furthermore, the single dose corresponds to at least two to three time times higher biological effective dose than conventional fractionated external beam radiotherapy. Another potential advantage is the prevention of tumor cell proliferation during the post-operative period prior to start of adjuvant radiotherapy.

In this study, the investigators will use low energy x-rays (photons) to treat spine lesions during kyphoplasty. The IORT device used will be the Intrabeam®, which is a miniature X-ray generator that produces low-energy X-rays: electrons are accelerated with a voltage of 30-50 kilovolts (kV) and hit a gold target at the tip of the drift tube. At this point the low-energy radiation is generated and emitted isotropically, similar to a point source. Due to its sharp dose fall off, minimal radiation protection is required in the operating room. The ultimate goal is to treat tumor cells with optimal sparing of spinal cord. (Please refer to Section 2.4 for more information on Intrabeam®).

Researchers at the University Medical Center in Mannheim, Germany completed a phase I trial assessing the tolerability of the Kypho-IORT procedure. Investigators reported their experience on performing the Kypho-IORT procedure in 18 patients (twenty-one vertebral lesions) with unstable or painful spinal metastases. The researchers used Intrabeam® to deliver 8Gy at 5mm distance from the spinal applicator surface using 50kV x-rays. The median age was 63 years and median follow up was 4.5 months (range, 1-10 months).

The procedure was well-tolerated. The median surgical time was 70 minutes (range, 53-173 minutes), which included radiation delivery time of approximately two minutes. Of the 21 vertebral lesions, 18 were treated successfully (86%). During the procedure, 78% of patients were noted to have asymptomatic paravertebral para-methoxymethamphetamine (PMMA) cement leakage. None of the treated patients had delayed wound healing, spinal or nerve root compression, paresthesia, new neurological deficit, or skin toxicity.

In terms of pain relief, the median visual analog pain score (VAS) was 5 prior to procedure. The VAS decreased to 2.5 on the first post-procedure day. At six weeks, 12 of the 18 patients were available to be evaluated and reported a median VAS score of 0/10. 67% of the patients required analgesic medication for pain relief prior to procedure, but decreased to just 30% at six weeks. Furthermore, imaging studies were available for 15 of the 18 patients, revealing 93% (14/15) patients had stable disease. Only one patient had progressive disease based on radiographic evidence, but this patient did not require any additional intervention.

INTRABEAM:

The Intrabeam® machine delivers low energy 50-kV photons directly to a target volume. The device generates electrons and then, accelerates them in a sealed vacuum probe (drift tube, measures 10 cm long and 3.2 mm in outer diameter). This drift tube, located within the x-ray spectrometer (XRS) unit, incorporates a gold target on the inside surface of its tip. When the accelerated electrons collide with the gold target at the end of the drift tube, photons are generated and dispersed in an isotropic dose distribution. The X-ray source itself is mounted on a balanced floor stand with six degrees of freedom to provide various treatment positions. The Intrabeam® system is calibrated for quality assurance prior to each treatment.

For the Kypho-IORT procedure, specially designed spinal applicator tip is used. This sterile applicator tip consists of a plastic head, which attaches to the drift tube and is then, placed inside a stainless steel tube (metallic sleeve). The applicator tip protects the drift tube from bending. The applicator is made of plastic in order to minimize the absorption and attenuation of the photons. Under fluoroscopic guidance, the applicator tip is guided though the metallic sleeves to the placed in mid-point/mid-plane of the vertebral lesion.

Due to the steep dose fall-off, a high dose to the vertebral lesion can be delivered, with maximum sparing of spinal cord. A radiation dose of 8 Gy at a distance of 5 mm from the applicator surface will be prescribed. This correlates to an approximate dose of 91 Gy at the applicator surface, 45 Gy at a distance of 1mm (from the applicator surface), 27Gy at 2mm, and 8Gy at 5mm. Further dose fall off is approximated: 2.4Gy at 10mm, 0.8Gy at 15mm, and 0.4Gy at 20mm. Assuming minimal distance of 15mm to the spinal cord, then, the spinal cord would receive less than 1Gy.

Study Design:

The combination of intraoperative radiotherapy with kyphoplasty will provide immediate vertebra stabilization, durable pain relief, and sterilization of tumor cells in a single outpatient procedure. To this date, this procedure has not been performed in the United States. The investigators plan to conduct a phase I trial of Kypho-IORT at the Loyola University Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic patients from solid tumor
* Estimated life expectancy of at least 3 months
* Age >= 50 years.
* Karnofsky Performance Status >= 70%
* Numeric Pain Intensity Score >= 3
* 10% or more loss of vertebrae height
* Adequate organ and marrow function as defined below:
* International normalized ratio (INR)/ prothrombin time (PT) within normal institutional limits
* leukocytes >= 3,000 microliter (mcL)
* Absolute neutrophil count >= 1,500 mcL
* Platelets >= 100,000 mcl
* Total bilirubin within normal institutional limits
* Abnormal aspartate transaminase (AST or SGOT) or alanine transaminase (ALT or SPGT)
* Abnormal creatinine
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Patients who have had prior external beam radiotherapy or surgery in the area of planned intervention
* Previous radiopharmaceuticals (i.e, Ra-222, Sr-90, etc) within 30 days of procedure
* Patients who are receiving systemic therapy (chemotherapy, hormonal, immunotherapy, bisphosphonates, etc) or other investigational agents are eligible if the systemic therapy can be safely held two weeks prior to procedure. These therapies may be resumed two weeks after the procedure
* Primary hematologic malignancies
* Patients with clinical or radiographic evidence of spinal cord or cauda equine compression or effacement
* Chronic vertebrae fracture of greater than 6 months or coexisting bilateral pedicle fracture
* Previous kyphoplasty in the same area
* Patients with severe spinal deformity requiring open reconstruction or extreme adiposity, in which determining placement of metal sleeve would be difficult by fluoroscopy (limited bone margin)
* History of allergic reactions attributed to compounds of similar composition to agents used for kyphoplasty
* Uncontrolled medical illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pre-menopausal female

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-12; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Pain | 52 weeks
  Patient will rate the severity of pain on a numeric 0-10 scale with higher scores indicating more severe pain. Pain assessment will be done at baseline, day of the procedure, and during follow up visits for up to 52 weeks.

SECONDARY OUTCOMES:
Tumor Response | 52 weeks
  Patients will be classified at week 52 as having (1) disappearance of the treated lesion (i.e., complete response), (2) at least 30% decrease in the diameter of the treated lesion (i.e., partial response), (3) at least 20% increase in the diameter of the treated lesion (i.e., progressive disease), or (4) Neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease (i.e., stable disease).

CONTACTS AND LOCATIONS:
Overall Officials: William Small, MD, Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

REFERENCES:
- [Background] Bartels RH, van der Linden YM, van der Graaf WT. Spinal extradural metastasis: review of current treatment options. CA Cancer J Clin. 2008 Jul-Aug;58(4):245-59. doi: 10.3322/CA.2007.0016. Epub 2008 Mar 19. PMID 18354080
- [Background] Ben-Josef E, Shamsa F, Williams AO, Porter AT. Radiotherapeutic management of osseous metastases: a survey of current patterns of care. Int J Radiat Oncol Biol Phys. 1998 Mar 1;40(4):915-21. doi: 10.1016/s0360-3016(97)00927-9. PMID 9531377
- [Background] Coleman RE. Metastatic bone disease: clinical features, pathophysiology and treatment strategies. Cancer Treat Rev. 2001 Jun;27(3):165-76. doi: 10.1053/ctrv.2000.0210. PMID 11417967
- [Background] Eck JC, Nachtigall D, Humphreys SC, Hodges SD. Comparison of vertebroplasty and balloon kyphoplasty for treatment of vertebral compression fractures: a meta-analysis of the literature. Spine J. 2008 May-Jun;8(3):488-97. doi: 10.1016/j.spinee.2007.04.004. Epub 2007 May 29. PMID 17588820
- [Background] Fourney DR, Schomer DF, Nader R, Chlan-Fourney J, Suki D, Ahrar K, Rhines LD, Gokaslan ZL. Percutaneous vertebroplasty and kyphoplasty for painful vertebral body fractures in cancer patients. J Neurosurg. 2003 Jan;98(1 Suppl):21-30. doi: 10.3171/spi.2003.98.1.0021. PMID 12546384
- [Background] Hage WD, Aboulafia AJ, Aboulafia DM. Incidence, location, and diagnostic evaluation of metastatic bone disease. Orthop Clin North Am. 2000 Oct;31(4):515-28, vii. doi: 10.1016/s0030-5898(05)70171-1. PMID 11043092
- [Background] Hartsell WF, Scott CB, Bruner DW, Scarantino CW, Ivker RA, Roach M 3rd, Suh JH, Demas WF, Movsas B, Petersen IA, Konski AA, Cleeland CS, Janjan NA, DeSilvio M. Randomized trial of short- versus long-course radiotherapy for palliation of painful bone metastases. J Natl Cancer Inst. 2005 Jun 1;97(11):798-804. doi: 10.1093/jnci/dji139. PMID 15928300
- [Background] Janjan NA. Radiation for bone metastases: conventional techniques and the role of systemic radiopharmaceuticals. Cancer. 1997 Oct 15;80(8 Suppl):1628-45. doi: 10.1002/(sici)1097-0142(19971015)80:8+3.3.co;2-l. PMID 9362430
- [Background] Kraus-Tiefenbacher U, Steil V, Bauer L, Melchert F, Wenz F. A novel mobile device for intraoperative radiotherapy (IORT). Onkologie. 2003 Dec;26(6):596-8. doi: 10.1159/000074158. No abstract available. PMID 14709937
- [Background] Krishnan MS, Epstein-Peterson Z, Chen YH, Tseng YD, Wright AA, Temel JS, Catalano P, Balboni TA. Predicting life expectancy in patients with metastatic cancer receiving palliative radiotherapy: the TEACHH model. Cancer. 2014 Jan 1;120(1):134-41. doi: 10.1002/cncr.28408. Epub 2013 Oct 2. PMID 24122413
- [Background] Li S, Peng Y, Weinhandl ED, Blaes AH, Cetin K, Chia VM, Stryker S, Pinzone JJ, Acquavella JF, Arneson TJ. Estimated number of prevalent cases of metastatic bone disease in the US adult population. Clin Epidemiol. 2012;4:87-93. doi: 10.2147/CLEP.S28339. Epub 2012 Apr 10. PMID 22570568
- [Background] Maranzano E, Latini P. Effectiveness of radiation therapy without surgery in metastatic spinal cord compression: final results from a prospective trial. Int J Radiat Oncol Biol Phys. 1995 Jul 15;32(4):959-67. doi: 10.1016/0360-3016(95)00572-g. PMID 7607970
- [Background] McCall T, Cole C, Dailey A. Vertebroplasty and kyphoplasty: a comparative review of efficacy and adverse events. Curr Rev Musculoskelet Med. 2008 Mar;1(1):17-23. doi: 10.1007/s12178-007-9013-0. PMID 19468894
- [Background] Reis T, Schneider F, Welzel G, Schmidt R, Bludau F, Obertacke U, Wenz F. Intraoperative radiotherapy during kyphoplasty for vertebral metastases (Kypho-IORT): first clinical results. Tumori. 2012 Jul-Aug;98(4):434-40. doi: 10.1177/030089161209800406. PMID 23052158
- [Background] Rose PS, Laufer I, Boland PJ, Hanover A, Bilsky MH, Yamada J, Lis E. Risk of fracture after single fraction image-guided intensity-modulated radiation therapy to spinal metastases. J Clin Oncol. 2009 Oct 20;27(30):5075-9. doi: 10.1200/JCO.2008.19.3508. Epub 2009 Sep 8. PMID 19738130
- [Background] Schneider F, Greineck F, Clausen S, Mai S, Obertacke U, Reis T, Wenz F. Development of a novel method for intraoperative radiotherapy during kyphoplasty for spinal metastases (Kypho-IORT). Int J Radiat Oncol Biol Phys. 2011 Nov 15;81(4):1114-9. doi: 10.1016/j.ijrobp.2010.07.1985. Epub 2010 Oct 8. PMID 20934272
- [Background] Wenz F, Schneider F, Neumaier C, Kraus-Tiefenbacher U, Reis T, Schmidt R, Obertacke U. Kypho-IORT--a novel approach of intraoperative radiotherapy during kyphoplasty for vertebral metastases. Radiat Oncol. 2010 Feb 11;5:11. doi: 10.1186/1748-717X-5-11. PMID 20149237
- [Background] Willett CG, Czito BG, Tyler DS. Intraoperative radiation therapy. J Clin Oncol. 2007 Mar 10;25(8):971-7. doi: 10.1200/JCO.2006.10.0255. PMID 17350946
- [Background] Wong DA, Fornasier VL, MacNab I. Spinal metastases: the obvious, the occult, and the impostors. Spine (Phila Pa 1976). 1990 Jan;15(1):1-4. PMID 2326692